CLINICAL TRIAL: NCT02348437
Title: Clinical Outcome After Repair of the Pronator Quadratus Muscle in Volar Locked Plating of the Distal Radius. A Randomised Clinical Trial.
Brief Title: Repair vs Non-repair of the Pronator Quadratus Muscle in Distal Radius Fractures. RCT.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Jesper Sonntag, MD, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PQ Project
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Radius Fractures; Colles' Fracture; Rupture of Muscle; Arm Injuries
Keywords: Pronator quadratus; Distal radius fracture; Repair; Volar plating; PRWE
MeSH Terms: conditions — Radius Fractures; Colles' Fracture; Arm Injuries; Wrist Fractures | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repair (Experimental): Repair of the pronator quadratus muscle
  Interventions: Procedure: Repair
- Non-repair (Active Comparator): Non-repair of the pronator quadratus muscle
  Interventions: Procedure: Non-repair

INTERVENTIONS:
Procedure: Repair — An on-going suture technique with minimum four stitches.
  Arms: Repair
Procedure: Non-repair — The PQ muscle will be placed so it covers the volar plate. No suture.
  Arms: Non-repair

SUMMARY:
The purpose of this study is to determine the functional outcome of repairing the pronator quadratus (PQ) muscle in subjects operated for a distal radius fracture (DRF) with volar locked plating.

DETAILED DESCRIPTION:
Fractures of the distal radius are common in the elderly. A frequent treatment of an unstable DRF is surgery with volar plating using the modified Henry's approach. In some cases the fracture mechanism has injured the PQ muscle and subsequent reconstruction of the muscle can be difficult. When the PQ muscle is not injured the plate is fixated through a radial and distal release of the PQ muscle and resuture/repair of the PQ muscle is attempted by most surgeons.

The clinical relevance of repairing the PQ muscle has not previously been investigated in a randomised clinical trial and we hypothesise that there is no difference in functional outcome whether the PQ muscle is repaired or not.

ELIGIBILITY:
Inclusion criteria:

* patients over 18 years.
* patients with an unstable DRF AO type 23 A2, A3, C1, C2 or C3 elected for surgery with volar plating. Unstable is defined as one of the following: 1) More than 10 degrees dorsal angulation of radius' joint surface in lateral plane measured from an orthogonal axis through radius. 2) Ulnar variance more than 2 mm. 3) Fracture line involving joint surface with more than 2 mm dislocation. 4) Incongruence of the DRJ.
* patients that can undergo the surgery in plexus brachialis block (so the operation can be performed in the outpatient department).
* patients with the ability to read and understand Danish.

Exclusion criteria:

* patients with an open fracture.
* patients with a neurologic disorder affecting the fractured upper extremity.
* patients with a history of fracture to the same wrist.
* patients with dementia, substance abuse or severe psychiatric disorder.
* patients who do not agree to be randomised.
* patients unable to continue follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 12 months

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) | 2 weeks, 5 weeks, 3 months, 6 months
Disabilities of the Arm, Shoulder and Hand (DASH) | 2 weeks, 5 weeks, 3 months, 6 months, 12 months
Pronation strength | 5 weeks, 3 months, 6 months, 12 months
Grip strength | 5 weeks, 3 months, 6 months, 12 months
Range of motion: supination/pronation | 2 weeks, 5 weeks, 3 months, 6 months, 12 months
Operation time | day 0
Ultra sonic examination (Examination of tendons and PQ muscle) | 3 months
  Examination of tendons and PQ muscle
Complications (Tendon rupture and Tendinitis) | 2 weeks, 5 weeks, 3 months, 6 months, 12 months
  Tendon rupture and Tendinitis

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonntag, MD, Principal Investigator — Nordsjaellands Hospital Hilleroed, Unit of Orthopaedic Surgery, Dyrehavevej 29, 3400 Hilleroed. Denmark
Locations (1):
- Nordsjaellands Hospital Hilleroed, Unit of Orthopaedic Surgery, Hilleroed, Denmark